CLINICAL TRIAL: NCT02103426
Title: A Phase 1, Single-Blind, Parallel-Group, Pharmacokinetic and Immunogenicity Study With ASP0113 in CMV-Seropositive and CMV-Seronegative Healthy Subjects and CMV-Seronegative Dialysis Patients
Brief Title: An Evaluation of a Cytomegalovirus (CMV) Vaccine (ASP0113) in CMV-Seropositive and CMV-Seronegative Healthy Subjects and CMV-Seronegative Dialysis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Vical (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0113-CL-0004
Record Dates: First submitted 2014-04-01; First posted 2014-04-03 (Estimated); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Dialysis; Healthy Subjects; Cytomegalovirus Infection
Keywords: Cytomegalovirus; ASP0113; CMV-seropositive; Healthy subjects; CMV-seronegative; Dialysis
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (10):
- Part 1: ASP0113 CMV-seropositive healthy cohort (Experimental): 5 mg single dose IM injection
  Interventions: Drug: ASP0113
- Part 1: ASP0113 CMV-seronegative healthy cohort (Experimental): 5 mg single dose IM injection
  Interventions: Drug: ASP0113
- Part 1: Placebo CMV-seropositive healthy cohort (Placebo Comparator): single dose IM injection
  Interventions: Drug: Placebo
- Part 1: Placebo CMV-seronegative healthy cohort (Placebo Comparator): single dose IM injection
  Interventions: Drug: Placebo
- Part 2: ASP0113 CMV-seropositive healthy cohort (Experimental): 4 IM injections of ASP0113
  Interventions: Drug: ASP0113
- Part 2: ASP0113 CMV-seronegative healthy cohort (Experimental): 4 IM injections of ASP0113
  Interventions: Drug: ASP0113
- Part 2: ASP0113 CMV-seronegative dialysis cohort (Experimental): 4 IM injections of ASP0113
  Interventions: Drug: ASP0113
- Part 2: Placebo CMV-seropositive healthy cohort (Placebo Comparator): 4 placebo IM injections
  Interventions: Drug: Placebo
- Part 2: Placebo CMV-seronegative healthy cohort (Placebo Comparator): 4 placebo IM injections
  Interventions: Drug: Placebo
- Part 2: Placebo CMV-seronegative dialysis cohort (Placebo Comparator): 4 placebo IM injections
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP0113 — intramuscular injection
  Arms: Part 1: ASP0113 CMV-seronegative healthy cohort; Part 1: ASP0113 CMV-seropositive healthy cohort; Part 2: ASP0113 CMV-seronegative dialysis cohort; Part 2: ASP0113 CMV-seronegative healthy cohort; Part 2: ASP0113 CMV-seropositive healthy cohort
Drug: Placebo — intramuscular injection
  Arms: Part 1: Placebo CMV-seronegative healthy cohort; Part 1: Placebo CMV-seropositive healthy cohort; Part 2: Placebo CMV-seronegative dialysis cohort; Part 2: Placebo CMV-seronegative healthy cohort; Part 2: Placebo CMV-seropositive healthy cohort

SUMMARY:
The purpose of the study is to determine whether ASP0113 (a CMV deoxyribonucleic acid [DNA] vaccine) can be detected in plasma after intramuscular (IM) injections, and to determine whether CMV-seropositive healthy volunteers, CMV-seronegative healthy volunteers, CMV-seronegative dialysis patients mount an immune response to the CMV proteins produced by the vaccine after repeated ASP0113 IM injection.

DETAILED DESCRIPTION:
Part 1 is open-label with no randomization, and Part 2 is single-blind and randomized. The purpose of Part 1 is to obtain pilot pharmacokinetic data so as to optimize pharmacokinetic sample collection times in Part 2.

ELIGIBILITY:
Inclusion Criteria:

Main Inclusion for Healthy Subjects:

* Body Mass Index (BMI) range of 18.5 - 35.0 kg/m2; weighs at least 50 kg at Screening.
* Female subject must not be lactating and must not be breast feeding within 3 months before Screening or during the study period and for 28 days after final injection.
* Female subject must not donate ova starting at Screening and throughout the study period and for 28 days after final injection.
* Highly likely to comply with the protocol and complete the study.
* Estimated creatinine clearance calculated using the Cockcroft-Gault equation of > 80 mL/min/1.73m2 (normal renal function).

Inclusion Criteria for Dialysis Patients:

* BMI range of 18.5 - 40.0 kg/m2; weighs at least 50 kg at Screening.
* Female subject must not be lactating and must not be breast feeding within 3 months before Screening or during the study period and for 30 days after final injection.
* Female subject must not donate ova starting at Screening and throughout the study period and for 28 days after final study drug administration.
* Must have adequate venous access.
* Highly likely to comply with the protocol and complete the study.
* Must currently be receiving hemodialysis treatment and for a period of at least 6 months prior to Screening.
* CMV-seronegative at Screening.

Exclusion Criteria:

Main Exclusion Healthy Subjects

* Female subject is pregnant at Screening.
* Any clinically significant history of allergic conditions (including drug allergies, asthma, eczema, or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies).
* Any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal (for healthy subjects only) and/or other major disease or malignancy (except non-metastatic basal or squamous cell carcinoma of the skin that has been treated successfully or cancer in situ of the cervix uteri that has been handled by local surgery).
* History or evidence of autoimmune diseases including systemic lupus erythematosus, rheumatoid arthritis, scleroderma, psoriasis, psoriatic arthritis and inflammatory bowel disease.
* Febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (non-cutaneous) infection within 1 week prior to day -14.
* Any of the liver function tests (LFT) (aspartate amino-transferase [AST] or alanine aminotransferase [ALT] alkaline phosphatase (ALP), gamma-glutamyl transferase [GGT], total bilirubin [TBil]) outside of normal limits at Screening.
* Mean pulse < 40 or > 90 beats per minute (bpm), mean systolic blood pressure (SBP) > 160 mmHg or mean diastolic blood pressure (DBP) > 90 mmHg taken in triplicate after the subject has been resting in a sitting position for at least 5 minutes at Screening.
* Positive serology test for hepatitis B surface antigen (HBsAg) or hepatitis core immunoglobulin M (HBc [IgM]) antibody, anti-hepatitis A virus (HAV) IgM or anti-human immunodeficiency virus type 1 and type 2 (HIV-1 and HIV-2) at Screening.
* Positive serology test for anti-hepatitis C virus (HCV) and a confirmatory positive reflex viral load test at Screening.
* Current/ active CMV infection as evidenced by positive CMV Polymerase chain reaction (PCR) plasma results at Screening.
* Any known or suspected hypersensitivity to ASP0113 or any components of the formulation used, including aminoglycosides as kanamycin is used during the manufacturing of the vaccine.
* Use of any prescribed or non-prescribed drugs, alternative and complementary medications, except for vitamins, contraceptives, hormone replacement therapy and occasional acetaminophen (to a maximum of 2 g/day), within 14 days prior to first injection with ASP0113.
* Vaccination with killed vaccines (including e.g., influenza and pneumococcal), or allergy treatment with antigen injections within 15 days prior to day -1.
* Vaccination with live attenuated vaccines within 30 days prior to day -1.
* Participated in any interventional clinical study or has been treated with any investigational drugs within 30 days or 5 half-lives, whichever is longer, prior to day 1.
* History of consuming more than 14 units of alcoholic beverages per week within 6 months prior to Screening or has a history of alcoholism or drug/chemical/substance abuse within past 2 years prior to Screening (Note: 1 unit = 12 ounces of beer, 4 ounces of wine or 1ounce of spirits/hard liquor).
* Positive test for alcohol or drugs of abuse at Screening or day -1.
* Significant blood loss, donation of 1 unit (450 mL) or more of blood or receipt of a transfusion of any blood, blood products or plasma within 90 days of day -1.
* Contraindication to an intramuscular (IM) injection.
* Employee of the Astellas Group or contract research organization (CRO) involved.

Exclusion Criteria for Dialysis Patients:

* Female subject is pregnant at Screening.
* Any clinically significant history of allergic conditions (including drug allergies, asthma, eczema, or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies).
* Any history or evidence of any unstable, clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, metabolic, pulmonary, neurologic, dermatologic, psychiatric and/or other major disease or malignancy.
* History of prior organ transplant, including a kidney, unless the transplant was unsuccessful and the subject is no longer receiving immunosuppressive therapy.
* History or evidence of autoimmune diseases including systemic lupus erythematosus, rheumatoid arthritis, scleroderma, psoriasis, psoriatic arthritis and inflammatory bowel disease or other disease which may require use of an immunosuppressant medication during the trial.
* Febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to day-14.
* Hemoglobin < 9 g/dL, TBil greater than the upper limit of normal (ULN), or an AST or ALT greater than 2 x the ULN at Screening. In such cases the assessment may be repeated once.
* Mean pulse < 40 or > 100 bpm or mean SBP > 180 mmHg; mean DBP > 100 mmHg taken in triplicate after the subject has been resting in a sitting position for at least 5 minutes at Screening.
* Positive serology test for HBsAg or HBc (IgM), anti HAV (IgM), anti-HIV-1 or anti-HIV-2 at Screening.
* Positive serology test for anti-HCV and a confirmatory positive reflex viral load test at Screening.
* Current/active CMV infection as evidenced by positive CMV PCR plasma results at Screening.
* Known or suspected hypersensitivity to ASP0113 or any components of the formulation used, including aminoglycosides as kanamycin is used during the manufacturing of the vaccine.
* Use of alternative and complementary medications except for vitamins, within 14 days prior to first injection with ASP0113.
* Subject has had use of any immunosuppressive drugs, including but not limited to, systemic corticosteroids within 14 days or 5 half-lives of initial injection, whichever is longer. History of topical or inhaled corticosteroid use should be discussed with the Medical Monitor for evaluation.
* Use of anticoagulants, including, but not limited to, vitamin K antagonists, heparin or its derivatives, low molecular weight heparin, factor X inhibitors or thrombin inhibitors within 5 half-lives of the first ASP0113 injection. Low dose anticoagulants used for prevention of deep vein thrombosis, prevention of fistula clotting, prevention of cardiovascular clotting, and heparin for use with dialysis procedure will be allowed after review and approval from the medical monitor.
* Vaccination with killed vaccines (including e.g., influenza and pneumococcal), or allergy treatment with antigen injections between the date of screening and day-1.
* Vaccination with live attenuated vaccines within 30 days prior to day-1.
* Participated in any interventional clinical study or treatment with any investigational drugs within 30 days or 5 half-lives, whichever is longer, prior to day 1.
* History of consuming more than 14 units of alcoholic beverages per week within 6 months prior to Screening or has a history of alcoholism or drug/chemical/substance abuse within past 2 years prior to Screening (Note: 1 unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits/hard liquor).
* Positive test for alcohol or drugs of abuse (non-prescribed) at Screening or day -1.
* Significant blood loss, donated 1 unit (450 mL) or more of blood or receipt of a transfusion of any blood, blood products or plasma within 90 days of day -14.
* Contraindication to an IM injection.
* Employee of the Astellas Group or CRO involved in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-12-30 (Actual); Primary Completion 2016-05-10 (Actual); Study Completion 2016-05-10 (Actual)

PRIMARY OUTCOMES:
ASP0113 plasmids pharmacokinetics in plasma: AUC (Part 1 and Part 2) | Day 1, 2, 3, 4, 5, 6, 7, 10, 14, 21 and 28 for Part 1; Day 1, 2, 3, 4, 5, 6, 7 and weeks 5, 9 and 25 for Part 2)
  Area under the curve (AUC)
ASP0113 plasmids pharmacokinetics in plasma: Cmax (Part 1 and Part 2) | Day 1, 2, 3, 4, 5, 6, 7, 10, 14, 21 and 28 for Part 1; Day 1, 2, 3, 4, 5, 6, 7 and weeks 5, 9 and 25 for Part 2
  Maximum Concentration (Cmax)
ASP0113 plasmids pharmacokinetics in plasma: Tmax (Part 1 and Part 2) | Day 1, 2, 3, 4, 5, 6, 7, 10, 14, 21 and 28 for Part 1; Day 1, 2, 3, 4, 5, 6, 7 and weeks 5, 9 and 25 for Part 2
  Time to maximum concentration (Tmax)
ASP0113 plasmids pharmacokinetics in plasma: Apparent clearance (Part 1 and Part 2) | Day 1, 2, 3, 4, 5, 6, 7, 10, 14, 21 and 28 for Part 1; Day 1, 2, 3, 4, 5, 6, 7 and weeks 5, 9 and 25 for Part 2
ASP0113 plasmids pharmacokinetics in plasma: apparent volume of distribution (Part 1 and Part 2) | Day 1, 2, 3, 4, 5, 6, 7, 10, 14, 21 and 28 for Part 1; Day 1, 2, 3, 4, 5, 6, 7 and weeks 5, 9 and 25 for Part 2
ASP0113 plasmids pharmacokinetics in plasma: half-life (Part 1 and Part 2) | Day 1, 2, 3, 4, 5, 6, 7, 10, 14, 21 and 28 for Part 1; Day 1, 2, 3, 4, 5, 6, 7 and weeks 5, 9 and 25 for Part 2
pp65 protein in white blood cells (WBCs) using pp65 antigenemia assay (Part 1 and Part 2) | Day 1, 2, 3, 4, 5, 6, 7, 10, 14, 21 , 28 for Part 1; Day 1, 10, 14, weeks 5, 7, 9, 11, 25 and 27 for Part 2
Immunogenicity: Relative units/ml of anti-gB antibodies in serum as detected by enzyme-linked immunosorbent assay (ELISA) (Part 2) | Day 1 and weeks 3, 5, 7, 9, 11, 25 and 27 (Part 2)
Immunogenicity: Number of pp65-specific Interferon (IFN)-gamma producing T-cells in isolated peripheral blood mononuclear cells (PBMCs) upon pp65 peptide stimulation as assayed by flow cytometry with intracellular cytokine staining (ICS) (Part 2) | Day 1 and weeks 3, 5, 7, 9, 11, 25 and 27 (Part 2)
Immunogenicity: Amount of IFN-gamma produced by CMV peptide-stimulated T-cells in whole blood using the QuantiFERON T-cell CMV assay (Part 2) | Day 1 and weeks 3, 5, 7, 9, 11, 25 and 27 (Part 2)
Safety assessed by clinical labs, vital signs, and adverse events including local and systemic reactogenicity | Up to Day 28 (Part 1), Up to 7 months (Part 2)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (4):
- United States (4):
  - Site US10009, Los Angeles, California
  - Site US10003, Orlando, Florida
  - Site US10001, Baltimore, Maryland
  - Site US10004, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=309